CLINICAL TRIAL: NCT04062851
Title: Routine Versus no Assessment of Gastric Residual Volumes in Very Low Birth Weight Infants Receiving Enteral Feeding Via Intermittent Feeding Tubes: A Randomized Controlled Trial.
Brief Title: Routine Versus no Assessment of Gastric Residual Volumes in Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AdventHealth (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1255832
Record Dates: First submitted 2019-04-09; First posted 2019-08-20 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Gastric Residual Volume; Preterm Infant; Feeding Disorder Neonatal
Keywords: gastric residuals, feeding, very low birth weight infants
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Intervention Model Description: Unblinded Single center Randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GRV group (No Intervention): Gastric residuals will be checked prior to feeds
- NO GRV group (Experimental): Gastric residuals will not be checked prior to feeds
  Interventions: Other: No Gastric residual volume monitoring

INTERVENTIONS:
Other: No Gastric residual volume monitoring — Gastric residual volumes will not be monitored
  Arms: NO GRV group

SUMMARY:
The practice of checking gastric residuals is not evidence based. The amount of gastric residual volume (GRV) does not correlate with either feeding intolerance or development of NEC. We hypothesize that not monitoring GRV in infants with birth weights < 1,250 g, and who are being fed intermittently by gastric tube, will result in earlier attainment of full feeding. This is an unblinded randomized controlled trial where GRV will not be checked routinely in the intervention group.

DETAILED DESCRIPTION:
The term "gastric residuals" in neonates refers to aspiration of gastric contents before each feeding in an infant receiving enteral feeding using an intermittent feeding tube. The presence of significant gastric residual volume (GRV) (Greater than 50% of the feeding volume) is a manifestation of delayed gastrointestinal maturation in a preterm neonate. The presence of GRV and its characteristics usually delays advancement of enteral feedings in premature infants because a large volume of undigested milk usually prompts the clinicians to hold the feeding.

Advancement of early enteral nutrition is delayed or discontinued for >24 hours in nearly 75% of all extremely preterm infants. This is despite clinical evidence showing that early establishment of enteral nutrition is associated with reductions in the severity of critical illness, and long-lasting benefits on linear growth and neurodevelopmental outcomes.

The magnitude and characteristics of GRV combined with specific findings based on abdominal examinations are usually considered by clinicians in decisions to continue with the scheduled enteral feeding plan. There are no studies to establish the normal volume of gastric residuals, its characteristics and whether routinely checking for them prior to each feed prevents necrotizing enterocolitis. A recent cohort study using retrospective controls showed that not monitoring GRV is associated with earlier attainment of full feeding in very low birth weight infants. Two small randomized studies conducted outside the United States and one study conducted in the United States showed no difference in outcomes when GRV are not checked routinely in preterm infants. These studies have several drawbacks and the practice of checking GRV continues.

Study Objectives

Primary Objective/Aim/Goal/Hypothesis

The primary objective of this study is to demonstrate that not monitoring GRV in infants with birth weights < 1,250 g, and who are being fed intermittently by gastric tube, will result in earlier attainment of full feeding.

Hypothesis:

In preterm infants, changing the clinical practice from routine gastric residuals evaluation to no aspiration for gastric residuals will decrease the number of days to reach full enteral feeds.

Secondary Objective/Aim/Goal/Hypothesis

A secondary objective is to show that there will be no difference in the incidence of NEC (necrotizing enterocolitis) in the experimental vs the control group.

Sample Size Determination

Our NICU database shows that for infants <1,250 g the days to full feeding was 16.4 ±7.3 days. To detect a relative decrease of 20% in the experimental group will require 73 infants in each group with an alpha of 0.05 and a power of 0.8.

Statistical Analysis Plan

Primary Objective Analysis

The primary outcome analysis is the number of days to reach full feeding volume, defined as volume > 120 ml/kg/d. This time will be compared between the two groups using analysis of variance.

Secondary Objective Analysis

Secondary analysis will be focused the frequency of feeding interruptions, incidences of NEC between the two groups using analysis of variance.

ELIGIBILITY:
Inclusion Criteria:

1. Birth weight ≤1250g
2. Gestational age of < 33 weeks
3. Expected to receive feeds via gastric tubes

Exclusion Criteria:

1. Death expected within 72 hours of birth
2. Major chromosomal or congenital anomaly
3. Major GI anomaly such as gastroschisis, spontaneous perforation etc.

Ages: 2 Hours to 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2019-05-03 (Actual); Primary Completion 2021-07-26 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Days to reach full enteral feeds | 1 month after enrollment
  Days to reach enteral feeding volume of 120ml/kg/day

SECONDARY OUTCOMES:
Necrotizing enterocolitis | Until hospital discharge, an average of 2-6 months
  Stage 2 NEC and higher grade
weight gain | 4 weeks chronological age and 36 weeks corrected gestation
  Weight gain velocity in gm/kg/d
frequency of feeding interruptions | Until full feeds are reached, usually between 2 weeks - 2 months
  Number of timed feeds are withheld

CONTACTS AND LOCATIONS:
Overall Officials: Narendra Dereddy, MD, Principal Investigator — AdventHealth
Locations (1):
- AdventHealth, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Li YF, Lin HC, Torrazza RM, Parker L, Talaga E, Neu J. Gastric residual evaluation in preterm neonates: a useful monitoring technique or a hindrance? Pediatr Neonatol. 2014 Oct;55(5):335-40. doi: 10.1016/j.pedneo.2014.02.008. Epub 2014 Aug 14. PMID 25129325
- [Result] Torrazza RM, Parker LA, Li Y, Talaga E, Shuster J, Neu J. The value of routine evaluation of gastric residuals in very low birth weight infants. J Perinatol. 2015 Jan;35(1):57-60. doi: 10.1038/jp.2014.147. Epub 2014 Aug 28. PMID 25166623
- [Result] Parker L, Torrazza RM, Li Y, Talaga E, Shuster J, Neu J. Aspiration and evaluation of gastric residuals in the neonatal intensive care unit: state of the science. J Perinat Neonatal Nurs. 2015 Jan-Mar;29(1):51-9; quiz E2. doi: 10.1097/JPN.0000000000000080. PMID 25633400